CLINICAL TRIAL: NCT03839797
Title: Adapting, Developing, And Testing An Evidence-Based Life Skills Training Approach For Sexual Assault Prevention
Brief Title: Cadet Healthy Personal Skills Intervention Trial
Acronym: CHiPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Promotion Associates, Inc. (Industry)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kenneth W Griffin, Senior Research Scientist, National Health Promotion Associates, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FAC20170050H
Record Dates: First submitted 2019-02-04; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Sexual Behavior; Skills, Social; Skills, Coping
MeSH Terms: conditions — Sexual Behavior; Social Skills

STUDY DESIGN:
Intervention Model Description: Half of the squadrons of incoming cadets were randomized to the CHiPS intervention, the other half were randomized to the control condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cadet Healthy Personal Skills (Experimental): Cadet Healthy Personal Skills
  Interventions: Behavioral: Cadet Healthy Personal Skills
- Standard Health Education (Active Comparator): Standard Health Education
  Interventions: Behavioral: Standard Health Education

INTERVENTIONS:
Behavioral: Cadet Healthy Personal Skills — 7.5 hour skills training group intervention
  Arms: Cadet Healthy Personal Skills
Behavioral: Standard Health Education — Standard Health Education
  Arms: Standard Health Education

SUMMARY:
The purpose of this study is to evaluate a new approach to sexual violence prevention by promoting healthy relationships and personal life skills among incoming Air Force cadets at the United States Air Force Academy.

DETAILED DESCRIPTION:
National Health Promotion Associates (NHPA) adapted the Botvin Life Skills Training (LST) program for incoming fourth class cadets at the United States Air Force Academy (USAFA). The resulting adaptation, called Cadet Healthy Personal Skills (CHiPS), provides cadets with the knowledge, attitudes, and skills to enhance their personal resilience, increase their potential for success, help them develop healthy and rewarding personal relationships, and reduce sexual harassment and assault. The CHiPS program includes ten units, spread across three blocks of content, and each block teaches cadets a range of life skills. All incoming fourth class cadets (N=1,203) were invited to participate in this study, beginning in the Summer of 2017, and of those, 1,098 cadets (91.3%) consented to participate in the trial.Twenty-five facilitators were trained to implement the newly adapted CHiPS program. Half of the incoming class [four Basic Cadet Training (BCT) squadrons] was assigned to receive the intervention, while the other half (four BCT squadrons) continued to receive standard trainings already in place at USAFA. All cadets completed a self-report survey at pretest, posttest, and at a 12-month follow-up

ELIGIBILITY:
Inclusion Criteria:

* incoming cadet at USAFA

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2017-08-05 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Self-reported sexual acts without consent | Past 1 year
  Three survey items assessed whether the participant was kissed or sexually touched without active consent, penetration or oral sex without active consent, or had sexual intercourse without consent and too intoxicated to resist.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth W Griffin, PhD, Principal Investigator — National Health Promotion Associates
Locations (1):
- National Health Promotion Associates, White Plains, New York, United States

REFERENCES:
- [Derived] Griffin KW, Williams C, Travis W, Tharp A. Prevention of Unwanted Sexual Contact Among Cadets at the United States Air Force Academy: A Brief Small-Group Intervention. Am J Public Health. 2021 Apr;111(4):672-674. doi: 10.2105/AJPH.2020.306050. Epub 2021 Jan 21. PMID 33476231